CLINICAL TRIAL: NCT01771757
Title: Measurement of Retinal Venous Pressure (Retinal Venous Pressure RVP) Under Conditions of Reduced Ambient Pressure and Oxygen Partial Pressure
Brief Title: Measurement of Retinal Venous Pressure Under Short-term Low-oxygen Environment
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: USB-2011-327
Record Dates: First submitted 2012-10-24; First posted 2013-01-18 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
Keywords: retinal venous pressure; reduced ambient pressure; oxygen partial pressure; short-term hypoxic changes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The hypothesis is that the pressure in the retinal veins increases under a short-term lack of oxygen and leads to a decreased blood circulation. On the basis of measurements in the hypobaric chamber this hypothesis should be verified.

DETAILED DESCRIPTION:
Conduct a pilot study to describe and quantify the retinal venous pressure (RVP) in healthy volunteers under conditions of controlled, reduced ambient and oxygen partial pressure in the pressure chamber of the Aeromedical Institute FAI in Dübendorf, Switzerland. Obtaining evidence of the adaptation behavior of the retinal vascular system in controlled, short-term hypoxic changes.

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* eye diseases
* systemic diseases
* term medication (except contraceptives)
* pregnancy
* allergies to the ingredients Alcain, Tropicamide and Phenylephrine
* blood pressure levels except standard (<60 /> 140 mmHg)
* oxygen saturation (SO2) <90%

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2011-12; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Retinal venous pressure | 1 hour
  Quantify the changes in the retinal venous pressure (RVP)

CONTACTS AND LOCATIONS:
Overall Officials: Josef Flammer, MD, Study Director — University of Basel, Dept. of Ophthalmology
Locations (1):
- University of Basel, Dept. of Ophthalmology, Basel, Switzerland